CLINICAL TRIAL: NCT04532255
Title: Periodontal Health Knowledge Among Patients With Fixed Orthodontic Appliance: A Hospital Based Cross-sectional Study
Brief Title: Periodontal Health Knowledge Among Patients With Fixed Orthodontic Appliance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Fekry Abbas El belkemy, Principal Investigator, Cairo University
Other Study IDs: PER 1-1-1
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a cross-sectional survey investigating the Periodontal health knowledge among patients with fixed orthodontic appliance attending the orthodontic department and the paid section faculty of dentistry Cairo University.

The faculty of Dentistry, Cairo University is an open public facility, a tertiary healthcare and a referral center.

DETAILED DESCRIPTION:
Dental patients will be recruited in a consecutive manner from orthodontic department faculty of dentistry Cairo University.

* Medical history will be taken, thorough oral examination will be done, and a full questionnaire will be filled for each patient.
* Full questionnaire will be filled, then full mouth periodontal examination and charting will be done for each patient.
* The questionnaire will be filled through a face-to-face personal interview with the patient using simple, short, easily comprehended questions.
* The interview questions will be prepared in English, translated into Arabic and then reverse translated by a certified translator to ensure accuracy.
* All the interviews done by the same investigator.
* Before the interview, the aim of the study will be explained to the patient and the patient's acceptance to participate in the survey will be received.
* Non-respondent patients or patients refusing to participate will be reported with the cause of their refusal.
* Conventional clinical examination will be held on a dental unit using the light of the unit, mirror and probe.
* Periodontal status will be evaluated including assessment of gingival index (GI), plaque index (PI), probing pocket depth (PPD) and number of teeth with gingival recession by using UNC 15 periodontal probe which is 15mm long probe with markings at each millimeter and color coded at 5th ,10th and 15th mm.
* The questionnaire which was applied in previous study will include the following:
* A series of questions related to demographic characteristics of the individuals; age, gender, duration of fixed orthodontic treatment, and the patient's current oral health behaviour (frequency and duration of tooth brushing, and auxiliary aids).
* Questions about periodontal knowledge of the individuals.
* Questions about awareness of patients toward the periodontal health.
* Questions related to subject's attitude toward orthodontic treatment and periodontal health.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age is 15-35 years old.
2. Patients with upper and lower fixed orthodontic appliances.
3. The duration of orthodontic treatment is 12 ±8 months.
4. All subjects were instructed for the need to properly clean the teeth after placing the appliance.
5. Provide informed consent

Exclusion Criteria:

1. Individuals with chronic systemic diseases such as diabetes, endocrine and haematological pathologies.
2. Patients having problem in opening their mouth or undergoing intermaxillary fixation where oral examination will not be possible.
3. Pregnant women.
4. Patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs.
5. Patients with congenital disorders or craniofacial anomalies such as cleft lip and palate and advanced (Sever) Periodontitis.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients with fixed orthodontic appliance attending the orthodontic department and the paid section faculty of dentistry Cairo University.
Sampling Method: Probability Sample
Enrollment: 314 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Periodontal health knowledge in patients receiving fixed orthodontic treatment. | An average of 1 year through study completion.
  will be assessed from Six questions about periodontal knowledge of the individuals and answers will be given in the form of multiple choices, with only one correct answer. These questions will be scored as 0 if the answer was in correct and as 1 if the answer was correct.

SECONDARY OUTCOMES:
The attitude and awareness toward orthodontic treatment and periodontal health. | An average of 1 year through study completion.
  will be assessed from Ten questions related to subject's awareness toward periodontal health that will be scored as 0 if the answer was "I don't know" and as 1 if the answer was "yes" or "no".
  The levels of awareness will be determined according to the scores and Ten questions related to subject's attitude toward orthodontic treatment and periodontal health that will be scored as 0 if the answer was negative and as 1 if the answer was positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medecine-CU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No